CLINICAL TRIAL: NCT00476333
Title: The Effect of Custom-Made Biomechanical Perturbation Platform on Kinetics, Kinematics and Electromyography in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 70/07
Record Dates: First submitted 2007-05-19; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-04

CONDITIONS: Healthy
Keywords: EMG; Kinetics; Kinematics; Perturbation; Footwear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: APOS biomechanical gait system

SUMMARY:
Introduction: Kinetic, kinematic and electromyographic activity of the lower limb have been shown to be influenced by various footwear-generated biomechanical manipulations (e.g. soles. Insoles, orthoses). A novel biomechanical device comprising four modular elements attached onto foot-worn platforms was recently developed. Each element can be individually calibrated (Position, convexity, height and resilience) to induce a specific biomechanical challenge.

Objectives: The aim of this study is to evaluate the influence of specific biomechanical challenges on Kinetics, kinematics and electromyographic activity of the lower limb.

Design: Prospective, case control Setting: Motion analyses will be conducted during level walking with (1) a three-dimensional motion analysis system and (2) ground reaction force analysis using force platforms (3) Electro-Myography system. Each subject will be examined in 16 different settings of the biomechanical system

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Similar anthorpometric profile (i.e. weight, shoe size, height, dominant leg)

Exclusion Criteria:

* Previous orthopedic, musculosceletal or neurological pathology

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nahum Halperin, MD, Principal Investigator — Asaf-Harofeh Medical Center
Locations (1):
- Technion Israel institute of technology, Biomechanical and bio-robotics division gait laboratory, Haifa, Israel